CLINICAL TRIAL: NCT02543463
Title: Comparison X3 Study Between Navi-THA and Non-navi-THA
Brief Title: Navigation With X3 vs Non-Navigation With X3 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCR-OR-1101v2
Record Dates: First submitted 2015-08-10; First posted 2015-09-07 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-09

CONDITIONS: Degenerative Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Navigation system (Other): Large diameter head with Trident X3 insert with Navigation system
  Interventions: Device: Trident X3 Insert with Navigation system
- Without Navigation system (Other): Large diameter head with Trident X3 insert with conventional instrumentation
  Interventions: Device: Trident X3 Insert with conventional instrumentation

INTERVENTIONS:
Device: Trident X3 Insert with Navigation system
  Arms: With Navigation system
Device: Trident X3 Insert with conventional instrumentation
  Arms: Without Navigation system

SUMMARY:
The purpose of this study is to compare the effect of the large head in THA with a navigation system and without a navigation system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is a candidate for a primary total hip arthroplasty (THA) with cementless acetabular and femoral components.
2. Patient who has a diagnosis of degenerative joint disease and no bacterial infectious disease.
3. Patient who is age 20 or over.
4. Patient who signed an Institutional Review Board (IRB)-approved, study specific Informed Patient Consent Form.
5. Patient who is willing to and able to comply with postoperative scheduled evaluations.

Exclusion Criteria:

1. Patient who has a bacterial infectious disease or has a high risk of a bacterial infection.
2. Patient who requires revision surgery of a previously implanted total hip arthroplasty.
3. Patient who is morbidly obese, defined as having a Body Mass Index (BMI) > 45.
4. Patient who is or may be pregnant female.
5. Patient who has neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
6. Patient with diagnosed systemic disease (i.e. Paget's disease, renal osteodystrophy).
7. Patient who is immunologically suppressed or receiving chronic steroids.
8. Patient who is judged ineligible with specific reason by primary doctor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) during surgery | intraoperative

SECONDARY OUTCOMES:
Measuring accuracy of the ROM during surgery | Intraoperative
  Measurement ROM precision of intraoperative
implantation accuracy | Intraoperative
  Measurement of the degree of stem anteversion, cup anteversion and cup abduction
Postoperative dislocation | From intraoperative to 1yr

CONTACTS AND LOCATIONS:
Overall Officials: Yasuyuki Inatsugu, Study Director — Stryker Japan
Locations (1):
- Osaka Rosai Hospital, Osaka, Osaka, Japan